CLINICAL TRIAL: NCT00730080
Title: Effects of Sapropterin on Brain and Cognition in Individuals With Phenylketonuria
Brief Title: Sapropterin in Individuals With Phenylketonuria
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: BioMarin Pharmaceutical (Industry); University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: PKU/Kuvan/White- 201104287
Record Dates: First submitted 2008-08-01; First posted 2008-08-08 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Phenylketonuria
Keywords: phenylketonuria; sapropterin; Kuvan; cognition; executive abilities; brain
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sapropterin (Kuvan): Individuals with phenylketonuria (PKU) who are beginning treatment with sapropterin.
  Interventions: Drug: Sapropterin (Kuvan)
- Control: Healthy individuals without phenylketonuria (PKU).

INTERVENTIONS:
Drug: Sapropterin (Kuvan) — 20mg/kg/day taken once daily or as otherwise prescribed by physician as standard care.
  Other Names: Kuvan
  Groups: Sapropterin (Kuvan)

SUMMARY:
Investigators at Washington University will examine the effects of sapropterin (Kuvan) on brain and cognition in individuals with phenylketonuria (PKU) using neuropsychological and neuroimaging procedures. Sapropterin is a medication developed by BioMarin Pharmaceutical Inc. that is approved by the FDA for treatment of patients with PKU to reduce phenylalanine (Phe) levels. Patients beginning treatment with sapropterin as standard clinical care will be enrolled in the study. As a first step, patients with PKU will receive baseline neuropsychological and neuroimaging evaluations 1 day prior to beginning treatment with sapropterin. Screening for response to sapropterin will occur over 4 weeks. At the end of 4 weeks, response to sapropterin will be reviewed. Patients with a reduction of ≥ 20% in blood Phe (i.e., responders) will receive follow-up neuropsychological and neuroimaging evaluations after 6 months of treatment with sapropterin. Patients (both responders and nonresponders) will receive long-term follow-up neuropsychological and neuroimaging evaluations 3 to 5 years after initial enrollment in the study.

The focus of neuropsychological testing will be executive abilities, as these abilities are particularly susceptible to disruption in individuals with PKU. We hypothesize that improvements in these abilities will occur following treatment with sapropterin. For neuroimaging assessments, structural magnetic resonance imaging (MRI) will permit evaluation of changes in the structure and volume of the gray and white matter of the brain, whereas diffusion tensor imaging (DTI) will permit evaluation of microstructural white matter integrity.

DETAILED DESCRIPTION:
Investigators at Washington University will examine the effects of sapropterin (Kuvan) on brain and cognition in individuals with phenylketonuria (PKU) using neuropsychological and neuroimaging procedures. Sapropterin is a medication developed by BioMarin Pharmaceutical Inc. that is approved by the FDA for treatment of patients with PKU to reduce phenylalanine (Phe) levels. Patients beginning treatment with sapropterin as standard clinical care will be enrolled. As a first step, patients with PKU who are ≥ 6 years of age will receive baseline neuropsychological and neuroimaging evaluations 1 day prior to beginning their treatment with sapropterin. Screening for response to sapropterin (20mg/kg/day) will then occur over 4 weeks as standard care for enrolled patients. At the end of 4 weeks, response to sapropterin will be reviewed. Patients with a reduction of ≥ 20% in blood Phe (i.e., responders) will receive follow-up neuropsychological and neuroimaging evaluations after 6 months of treatment with sapropterin. Patients (both responders and nonresponders) will receive long-term follow-up neuropsychological and neuroimaging evaluations 3 to 5 years after initial enrollment in the study.

A matched control group of healthy individuals without PKU will receive baseline and follow-up neuropsychological and neuroimaging evaluations for comparison purposes and to control for possible practice effects in repeated neuropsychological testing.

The focus of neuropsychological testing will be executive abilities, as these abilities are particularly susceptible to disruption in individuals with PKU. Specifically, the focus of neuropsychological assessment will be working memory, strategic processing, and inhibitory control, as our research group has shown that each of these executive abilities is impaired in individuals with PKU. (White, D. 2001 Neuropsychol.)(White, D. 2002 J. Int. Neuropsychol. Soc.)(Christ, S. 2006 Dev. Neuropsychol.) We hypothesize that improvements in these abilities will occur following treatment with sapropterin.

For neuroimaging assessments, both structural magnetic resonance imaging (MRI) and diffusion tensor imaging (DTI; mean diffusivity and fractional anisotropy) will be used. Structural MRI will permit evaluation of changes in the structure and volume of the gray and white matter of the brain. DTI will permit evaluation of microstructural white matter integrity. Brain abnormalities have been noted in individuals with PKU, and using DTI our research group recently identified abnormalities in the integrity of white matter in early and continuously treated individuals with PKU.

The primary objectives of the proposed study are two-fold. First, we will determine whether cognition (particularly executive abilities) improves in patients with PKU who have been treated with sapropterin. Second, we will determine whether the integrity of the brain improves in patients with PKU who have been treated with sapropterin. In addition, the interrelationships between changes in cognition and brain will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent or assent.
* Willing and able to comply with study procedures.
* Greater than or equal to 6 years of age.
* For phenylketonuria,intention of physician to prescribe sapropoterin.
* For phenylketonuria,phenylalanine level greater than or equal to 450μmol/L.
* For phenylketonuria, negative pregnancy test if of childbearing potential.
* For phenylketonuria, willing to use contraception if sexually active.

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during study.
* Use of investigational product less than 30 days prior to or during study.
* Concurrent condition that could interfere with participation or safety.
* Any condition creating high risk of poor compliance with study.
* Perceived to be unreliable or unavailable for study.
* Use of L-Dopa, methotrexate, or other drugs that inhibit folate metabolism.
* For phenylketonuria, known hypersensitivity to sapropterin or excipients.

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primary care clinic for phenylketonuria. St. Louis community for control.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
diffusion tensor imaging of the brain | baseline & follow-ups
  assesses functional white matter integrity

SECONDARY OUTCOMES:
n-back task | baseline & follow-ups
  assesses working memory
recognition span task | baseline & follow-ups
  assesses working memory
list learning task | baseline & follow-ups
  assesses strategic processing
verbal fluency task | baseline & follow-ups
  assesses strategic processing
go/no-go task | baseline & follow-ups
  assesses inhibitory control
stimulus-response compatibility task | baseline & follow-ups
  assesses inhibitory control
structural magnetic resonance imaging of the brain | baseline & follow-ups
  assesses structural brain integrity
Wechsler Abbreviated Scale of Intelligence | baseline & follow-ups
  assesses general intellectual ability

CONTACTS AND LOCATIONS:
Overall Officials: Desiree White, Ph.D., Principal Investigator — Washington University School of Medicine; Dorothy K. Grange, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] White DA, Nortz MJ, Mandernach T, Huntington K, Steiner RD. Deficits in memory strategy use related to prefrontal dysfunction during early development: evidence from children with phenylketonuria. Neuropsychology. 2001 Apr;15(2):221-9. doi: 10.1037//0894-4105.15.2.221. PMID 11324865
- [Background] White DA, Nortz MJ, Mandernach T, Huntington K, Steiner RD. Age-related working memory impairments in children with prefrontal dysfunction associated with phenylketonuria. J Int Neuropsychol Soc. 2002 Jan;8(1):1-11. PMID 11843066
- [Background] Christ SE, Steiner RD, Grange DK, Abrams RA, White DA. Inhibitory control in children with phenylketonuria. Dev Neuropsychol. 2006;30(3):845-64. doi: 10.1207/s15326942dn3003_5. PMID 17083296
- [Background] Araujo GC, Christ SE, Steiner RD, Grange DK, Nardos B, McKinstry RC, White DA. Response monitoring in children with phenylketonuria. Neuropsychology. 2009 Jan;23(1):130-4. doi: 10.1037/a0013488. PMID 19210041
- [Background] Christ SE, Huijbregts SC, de Sonneville LM, White DA. Executive function in early-treated phenylketonuria: profile and underlying mechanisms. Mol Genet Metab. 2010;99 Suppl 1:S22-32. doi: 10.1016/j.ymgme.2009.10.007. PMID 20123466
- [Background] White DA, Connor LT, Nardos B, Shimony JS, Archer R, Snyder AZ, Moinuddin A, Grange DK, Steiner RD, McKinstry RC. Age-related decline in the microstructural integrity of white matter in children with early- and continuously-treated PKU: a DTI study of the corpus callosum. Mol Genet Metab. 2010;99 Suppl 1(0 1):S41-6. doi: 10.1016/j.ymgme.2009.09.016. PMID 20123469
- [Background] Banerjee P, Grange DK, Steiner RD, White DA. Executive strategic processing during verbal fluency performance in children with phenylketonuria. Child Neuropsychol. 2011;17(2):105-17. doi: 10.1080/09297049.2010.525502. Epub 2010 Dec 7. PMID 21140312
- [Background] Janos AL, Grange DK, Steiner RD, White DA. Processing speed and executive abilities in children with phenylketonuria. Neuropsychology. 2012 Nov;26(6):735-43. doi: 10.1037/a0029419. Epub 2012 Aug 6. PMID 22866986
- [Result] Bodner KE, Aldridge K, Moffitt AJ, Peck D, White DA, Christ SE. A volumetric study of basal ganglia structures in individuals with early-treated phenylketonuria. Mol Genet Metab. 2012 Nov;107(3):302-7. doi: 10.1016/j.ymgme.2012.08.007. Epub 2012 Aug 18. PMID 23006929
- [Result] Antenor-Dorsey JA, Hershey T, Rutlin J, Shimony JS, McKinstry RC, Grange DK, Christ SE, White DA. White matter integrity and executive abilities in individuals with phenylketonuria. Mol Genet Metab. 2013 Jun;109(2):125-31. doi: 10.1016/j.ymgme.2013.03.020. Epub 2013 Apr 6. PMID 23608077
- [Result] Peng H, Peck D, White DA, Christ SE. Tract-based evaluation of white matter damage in individuals with early-treated phenylketonuria. J Inherit Metab Dis. 2014 Mar;37(2):237-43. doi: 10.1007/s10545-013-9650-y. Epub 2013 Sep 17. PMID 24043380
- [Result] White DA, Antenor-Dorsey JA, Grange DK, Hershey T, Rutlin J, Shimony JS, McKinstry RC, Christ SE. White matter integrity and executive abilities following treatment with tetrahydrobiopterin (BH4) in individuals with phenylketonuria. Mol Genet Metab. 2013 Nov;110(3):213-7. doi: 10.1016/j.ymgme.2013.07.010. Epub 2013 Jul 19. PMID 23928118